CLINICAL TRIAL: NCT00607984
Title: High Dose Thiotepa and Melphalan With Autologous Hematopoietic Stem Cell Transplant in Children and Adolescents With Solid Tumors
Brief Title: Administration of High Dose Thiotepa and Melphalan With Autologous Hematopoietic Stem Cell Transplant in Children and Adolescents With Solid Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Jerry Stein MD, Schneider Children's Medical Center of Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3990
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2008-01

CONDITIONS: Central Nervous System Tumors; Tumors
Keywords: thiotepa; melphalan; brain tumor; tumors of central nervous system and other solid tumors
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single (Experimental)
  Interventions: Drug: thiotepa melphalan

INTERVENTIONS:
Drug: thiotepa melphalan — thiotepa 900 mg per meter squared total, on days -11,-10,-4,-3 melphalan 140 mg per meter squared total on days -11,-10,-4,-3 autologous stem cell transplant in day 0

SUMMARY:
The prognosis of children and adolescents with high risk tumors of the central nervous system and other miscellaneous solid tumors is poor despite modern treatment protocols. Frequently, physicians suggest additional therapy with high dose chemotherapy after a good initial response to standard doses of treatment has been obtained, so as to reduce the chance that the tumor will recur. We propose a regimen of high dose thiotepa and melphalan followed by rescue of the patient's previously stored hematopoietic (blood manufacturing) system with blood stem cells. The aim of this study is to prove that this therapy is tolerable in children and adolescents, that it results in tolerable levels of toxicity, and that it improves the survival of this group of children as compared to standard therapy given in the past

DETAILED DESCRIPTION:
Despite progress in the treatment of children and adolescents suffering from solid tumors and tumors of the CNS, patients with metastatic disease (or with disease with other high risk features) continue to suffer from relapse when treated with standard chemotherapy protocols. In these patients, high-dose chemotherapy (HDC) followed by autologous stem cell transplantation (ASCT) has been proposed as consolidation therapy in this high-risk population.

The paradigm for successfully utilization of autologous stem cell transplantation is childhood neuroblastoma. A large, well performed, randomized study in children with high risk neuroblastoma showed that application of autologous stem cell transplant can lead to improved disease free and overall survival, effects that were further augmented by the administration of biological agents with specific activity against this tumor. Smaller non-controlled studies and case series have shown that ASCT is feasible in children with solid tumors or with tumors of the central nervous system. Despite the many reports in the literature, there is little agreement among investigators as to the ideal combination of chemotherapeutic agents that should be included in the high dose chemotherapy regimen administered prior to ASCT for these patients. The choice of agents in these protocols is dictated by the use of drugs whose dose limiting toxicity is hematopoietic, a concern that is obviated by the subsequent infusion of autologous stem cells. As such, the majority of HDC protocols exploit the steep dose response curve of alkylating agents, where administration of high doses had usually been limited by fear of inducing permanent myeloablation.

A major limitation of many HDC protocols is that many of the alkylating agents that are used have already been utilized in front line protocols. A further problem in the design of HDC protocols that is unique to patients suffering from CNS tumors, is that the administered agents must traverse the blood brain barrier (BBB) in order to reach the site of the tumor.

A major breakthrough in the the application of HDC in children nwith CNS tumors occurred with the use of Thiotepa, a highly myeloablative bifunctional alkylating agent that partitions equally across the BBB. Thiotepa is now a mainstay of all HDC protocols for children with CNS tumors.

Hara et al. pioneered a novel combination of Thiotepa with Melpahlan, also an alkylating agent, in the treatment of children with a variety of solid tumors. They catalogued the toxicity of this protocol, and suggested a dose level of each drug in the combination that led to toxicity levels of grade ≤3. Of note, in the Hara series, some patients also received high dose Busulfan.

We piloted the Hara protocol in our center on 14 patients and found that the dose levels suggested in their study were not tolerated well by children in our center. We decided to modify the Hara protocol by reducing the doses of both Thiotepa and Melphalan to reduce the incidence of severe gastrointestinal toxicity that our patients experienced. In addition, after two patients succumbed to fulminant gram positive infections on the original protocol, we instituted the empiric administration of Vancomycin for primary treatment of febrile neutropenia in these patients, pending the results of blood cultures. We also decided to restrict admission to the protocol to patients with minimal amounts of residual disease as measured by MRI / CT scan or biochemical markers prior to transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-21 years
* CNS tumors, hepatic tumors and other solid tumors that are chemosensitive
* Minimal disease as determined by either radiological studies or biochemical markers (as determined by treating physician).
* Consent of patient or surrogate.

Exclusion Criteria:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No known HIV or AIDS infection
* No active bacterial, fungal, or viral infection
* No medical condition that would preclude study treatment
* Positive pregnancy test or failure to use contraceptives.
* Creatinine >1.5 times limit of normal for age
* SGOT or SGPT more than 3 times normal.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-06; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
survival | 10 yeaer follow up

SECONDARY OUTCOMES:
toxicity | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Stein, MD, Principal Investigator — Schneider Children's Medical Center, Israel
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel